CLINICAL TRIAL: NCT00386152
Title: A Randomized, Open-Label, Comparative Study of Epoetin Alfa (PROCRIT) 80,000 Units or 120,000 Units Q3W (Every 3 Weeks) Versus Darbepoetin Alfa (ARANESP) 500 Mcg Q3W in Anemic Cancer Subjects Receiving Chemotherapy
Brief Title: A Study Comparing Two Different PROCRIT Doses to a Dose of ARANESP in Anemic Cancer Patients Receiving Chemotherapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: No safety signals were noted. The study was stopped because it was no longer consistent with the company's scientific and strategic focus.
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: Ortho Biotech Clinical Affairs, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR012985; EPOANE2007 (Other: Johnson & Johnson Pharmaceutical Research and Development, L.L.C.)
Record Dates: First submitted 2006-10-06; First posted 2006-10-11 (Estimated); Results first posted 2009-06-01 (Estimated); Last update posted 2013-07-19 (Estimated); Status verified 2013-07

CONDITIONS: Neoplasms; Anemia; Cancer
Keywords: Anemia; Cancer; Chemotherapy-Induced Anemia; Epoetin alfa; Darbepoetin alfa
MeSH Terms: conditions — Neoplasms; Anemia | interventions — Epoetin Alfa; Darbepoetin alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- epoetin alfa (120,000 Units) (Experimental): epoetin alfa (PROCRIT) 120,000 Units injected subcutaneously once every 3 weeks for up to 13 weeks
  Interventions: Drug: epoetin alfa
- epoetin alfa (80,000 Units) (Experimental): epoetin alfa (PROCRIT) 80,000 Units injected subcutaneously once every 3 weeks for up to 13 weeks
  Interventions: Drug: epoetin alfa
- darbepoetin alfa (500 mcg) (Active Comparator): darbepoetin alfa (ARANESP) 500 mcg injected subcutaneously the skin once every 3 weeks for up to 13 weeks
  Interventions: Drug: darbepoetin alfa

INTERVENTIONS:
Drug: epoetin alfa — 80,000 Units and 120,000 Units of epoetin alfa (PROCRIT) injected subcutaneously once every 3 weeks for up to 13 weeks
  Other Names: PROCRIT
  Arms: epoetin alfa (120,000 Units); epoetin alfa (80,000 Units)
Drug: darbepoetin alfa — 500 mcg of darbepoetin alfa (ARANESP) injected subcutaneously the skin once every 3 weeks for up to 13 weeks
  Other Names: ARANESP
  Arms: darbepoetin alfa (500 mcg)

SUMMARY:
The purpose of this study is to compare hemoglobin response rates between two PROCRIT (epoetin alfa) doses and ARANESP (darbepoetin alfa) in anemic cancer patients receiving chemotherapy

DETAILED DESCRIPTION:
This is an open-label (both the physician and the patient know which treatment is being provided), multi-center study of up to 16 weeks duration in which 450 patients will be randomly assigned (patients are assigned to a specific study group by chance) to one of three treatment groups in a 1:1:1 ratio. Patients will receive PROCRIT (epoetin alfa) 80,000 Units injected subcutaneously (under the skin) once every three weeks or 120,000 Units injected under the skin once every three weeks or ARANESP (darbepoetin alfa) 500 mcg injected under the skin once every three weeks for up to 13 weeks. PROCRIT (epoetin alfa) 80,000 Units and 120,000 Units given once every three weeks are doses and schedules that are not approved for use in the United States and are under investigation, while the ARANESP dose and schedule are approved for use in the United States. Adult patients with specific types of cancer (confirmed non-myeloid malignancy) who are scheduled to receive cyclic chemotherapy for a minimum of 12 weeks during the study and who meet all other eligibility criteria will be enrolled. This study will be conducted in approximately 80 study sites located in the United States.

The study hypothesis is that a dosing regimen of PROCRIT (Epoetin alfa) 80,000 Units or 120,000 Units given once every three weeks is non-inferior to ARANESP 500 mcg given once every three weeks with respect to the mean hemoglobin (Hb) change from baseline to Study Week 7 in anemic cancer patients receiving chemotherapy. Hemoglobin levels will be monitored throughout the study on a weekly basis and before each drug dose is administered. Drug dosing will be adjusted (ie, held, reduced, resumed at a lower dose) as needed to maintain hemoglobin values within desired ranges.

The maximum dose of PROCRIT (Epoetin alfa) allowed in this study is 120,000 Units every three weeks (Q3W) and the maximum dose of ARANESP (darbepoetin) is 500 mcg Q3W.

Safety evaluations will be conducted throughout the study and will consist of assessment of laboratory tests, vital signs, physical examinations. The occurrence and severity of adverse events, including thrombovascular events will be evaluated throughout the study.Periodic data monitoring of the study by an external Independent Data Monitoring Committee (IDMC) will be performed. The main responsibility of the IDMC is to conduct ongoing monitoring of safety and to report any irregularities back to the Sponsor along with recommendations regarding continuation of the study. Each patient will be assigned to one of three dosing schedules. All schedules will be administered by way of subcutaneous (under the skin) injection once every three weeks over a period of 13 weeks. The three dosing schedules are as follows: PROCRIT (epoetin alfa) 80,000 Units, PROCRIT (epoetin alfa) 120,000 Units or ARANESP (darbepoetin alfa) 500 mcg

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of a non-myeloid malignancy
* Baseline hemoglobin (Hb) value of <= 11.0 g/dL unrelated to transfusion
* No Packed Red Blood Cell (PRBC) or platelet transfusions in the 28 days prior to randomization
* Scheduled to receive chemotherapy for a minimum of 12 weeks during the study
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0 - 2

Exclusion Criteria:

* No planned non-palliative radiation during the study
* No current anemia due to factors other than cancer/chemotherapy (eg, iron deficiency or gastrointestinal bleeding)
* No uncontrolled hypertension (defined as systolic pressure > 180 and/or a diastolic pressure > 100 mmHg while receiving antihypertension therapy)
* No history of Deep Venous Thrombosis (DVT) or Pulmonary Embolus (PE) within 12 months before study enrollment. Prior superficial thrombophlebitis is not an exclusion criterion
* No history of Cerebrovascular Accident (CVA), Transient Ischemic Attack (TIA), Acute Coronary Syndrome (ACS) including unstable angina and myocardial infarction with or without ST elevation, or other arterial thrombosis within 6 months before study enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 235 (Actual)
Dates: Start 2006-11; Primary Completion 2008-03 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (76):
- United States (76):
  - Glendale, Arizona
  - Jonesboro, Arkansas
  - Little Rock, Arkansas
  - Anaheim, California
  - Bakersfield, California
  - Corona, California
  - Fountain Valley, California
  - Fullerton, California
  - Greenbrae, California
  - Irvine, California
  - La Jolla, California
  - La Verne, California
  - Lancaster, California
  - Long Beach, California
  - Los Angeles, California
  - Northridge, California
  - Orange, California
  - Rancho Mirage, California
  - Denver, Colorado
  - Norwich, Connecticut
  - Gainsville, Florida
  - Kissimmee, Florida
  - Lecanto, Florida
  - Pensacola, Florida
  - Athens, Georgia
  - Augusta, Georgia
  - Griffin, Georgia
  - Centralia, Illinois
  - Gurnee, Illinois
  - North Chicago, Illinois
  - Olympia Fields, Illinois
  - Park Ridge, Illinois
  - Springfield, Illinois
  - New Albany, Indiana
  - Hutchinson, Kansas
  - Kansas City, Kansas
  - Paducah, Kentucky
  - Baltimore, Maryland
  - Bethesda, Maryland
  - Worcester, Massachusetts
  - Free Soil, Michigan
  - Lansing, Michigan
  - Southfield, Michigan
  - Tupelo, Mississippi
  - Kansas City, Missouri
  - Omaha, Nebraska
  - Englewood, New Jersey
  - Clifton Springs, New York
  - Lake Success, New York
  - Asheville, North Carolina
  - Wilmington, North Carolina
  - Bismarck, North Dakota
  - Canton, Ohio
  - Lancaster, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pottsville, Pennsylvania
  - Aiken, South Carolina
  - Charleston, South Carolina
  - Mt. Pleasant, South Carolina
  - North Charleston, South Carolina
  - Sumter, South Carolina
  - Johnson City, Tennessee
  - Memphis, Tennessee
  - Bryan, Texas
  - El Paso, Texas
  - Galveston, Texas
  - Grapevine, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Tyler, Texas
  - Chesapeake, Virginia
  - Newport News, Virginia
  - Woodbridge, Virginia
  - Vancouver, Washington
  - Walla Walla, Washington
  - Morgantown, West Virginia

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Number of participants randomized:- epoetin alfa (80,000 Units): 77, epoetin alfa (120,000 Units): 80, darbepoetin alfa (500 mcg): 78; Number of participants treated:- epoetin alfa (80,000 Units): 75, epoetin alfa (120,000 Units): 77, darbepoetin alfa (500 mcg): 75.
Groups:
- Epoetin Alfa (80,000 Units): epoetin alfa (PROCRIT) 80,000 Units subcutaneous (SC) once every 3 weeks (Q3W) for up to 13 weeks
- Epoetin Alfa (120,000 Units): epoetin alfa (PROCRIT) 120,000 Units SC Q3W for up to 13 weeks
- Darbepoetin Alfa (500 Mcg): darbepoetin alfa (ARANESP) 500 mcg SC Q3W for up to 13 weeks
Period: Overall Study
Arm/Group | Epoetin Alfa (80,000 Units) | Epoetin Alfa (120,000 Units) | Darbepoetin Alfa (500 Mcg)
Started | 75 (number of subjects treated) | 77 (number of subjects treated) | 75 (number of subjects treated)
Completed | 31 | 37 | 42
Not Completed | 44 | 40 | 33
Not completed — Adverse Event | 6 | 5 | 4
Not completed — Chang from original chemo stratification | 4 | 5 | 6
Not completed — Death | 3 | 0 | 1
Not completed — Disease progression | 7 | 4 | 5
Not completed — Physician Decision | 13 | 10 | 4
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Completed chemotherapy | 4 | 5 | 1
Not completed — Protocol Violation | 3 | 5 | 2
Not completed — Withdrawal by Subject | 3 | 6 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Epoetin Alfa (80,000 Units) | Epoetin Alfa (120,000 Units) | Darbepoetin Alfa (500 Mcg) | Total
Number analyzed (Participants) | 77 | 80 | 78 | 235
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 36 | 34 | 41 | 111
  >=65 years | 41 | 46 | 37 | 124
Age Continuous [Mean (Standard Deviation); unit: years] | 65.05 (12.54) | 64.84 (11.66) | 63.00 (12.05) | 64.30 (12.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 57 | 52 | 150
  Male | 36 | 23 | 26 | 85
Chemotherapy Type [Number; unit: participants] — Randomization was stratified by chemotherapy type.
  participants
    Platinum | 29 | 32 | 30 | 91
    Non-Platinum | 48 | 48 | 48 | 144

OUTCOME MEASURES:

1. Secondary Outcome: Number of Patients Receiving at Least 1 Packed Red Blood Cell (PRBC) Transfusion During Study
Time Frame: up to 16 weeks
Population: modified intention-to-treat (mITT) population that includes the subjects who were randomized, received at least one dose of study medication, and had transfusion-unrelated Hb values obtained at baseline and at least one post baseline visit
Measure: Number; unit: participants
Arm/Group | Epoetin Alfa (80,000 Units) | Epoetin Alfa (120,000 Units) | Darbepoetin Alfa (500 Mcg)
Number analyzed (Participants) | 71 | 77 | 74
participants | 12 | 22 | 17

2. Primary Outcome: Hemoglobin (Hb) Change From Baseline to Study Week 7
Description: Baseline Hb was the Hb value that was consistent with the inclusion criteria and which was obtained within 72 hours of the first dose of study medication
Time Frame: Baseline (Week 1) and Week 7
Population: per-protocol (PP) population that includes a subset of the modified intent-to-treat (mITT) population with subjects who were randomized and received at least one dose of study medication, had transfusion-unrelated Hb values obtained at both baseline and Week 7, met inclusion and exclusion criteria, and had no major protocol violations up to Week 7
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Epoetin Alfa (80,000 Units) | Epoetin Alfa (120,000 Units) | Darbepoetin Alfa (500 Mcg)
Number analyzed (Participants) | 57 | 53 | 50
g/dL | 0.64 (1.30) | 0.40 (1.37) | 0.84 (1.28)

3. Secondary Outcome: Time to Achieve Hb >= 11 g/dL During Study
Time Frame: up to 16 weeks
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Epoetin Alfa (80,000 Units) | Epoetin Alfa (120,000 Units) | Darbepoetin Alfa (500 Mcg)
Number analyzed (Participants) | 71 | 77 | 74
days | 37 [29 to 50] | 44 [29 to 85] | 36 [29 to 44]

4. Secondary Outcome: Number of Patients (Hb >= 11 g/dL) During Study.
Time Frame: up to 16 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Epoetin Alfa (80,000 Units) | Epoetin Alfa (120,000 Units) | Darbepoetin Alfa (500 Mcg)
Number analyzed (Participants) | 71 | 77 | 74
participants | 51 | 48 | 56

ADVERSE EVENTS:
Arm/Group | Epoetin Alfa (80,000 Units) | Epoetin Alfa (120,000 Units) | Darbepoetin Alfa (500 Mcg)
Serious Adverse Events (participants affected / at risk) | 28/75 | 23/77 | 25/75
Other Adverse Events (participants affected / at risk) | 58/75 | 68/77 | 67/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Epoetin Alfa (80,000 Units) (N=75) | Epoetin Alfa (120,000 Units) (N=77) | Darbepoetin Alfa (500 Mcg) (N=75)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 1 | 2
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 2
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 3 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 1 | 1
Cardiopulmonary failure (Cardiac disorders) | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 0 | 0
Colonic obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0
Diabetic gastroparesis (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 2 | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0
Chest pain (General disorders) | 0 | 1 | 0
Systemic inflammatory response syndrome (General disorders) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0
Clostridial infection (Infections and infestations) | 1 | 0 | 0
Enterobacter sepsis (Infections and infestations) | 1 | 0 | 0
Klebsiella sepsis (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 4 | 1 | 2
Pneumonia fungal (Infections and infestations) | 0 | 1 | 0
Pneumonia herpes viral (Infections and infestations) | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 1 | 0
Sialoadenitis (Infections and infestations) | 0 | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 1 | 0 | 2
Urinary tract infection (Infections and infestations) | 0 | 2 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1
Compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Serum ferritin increased (Investigations) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 3 | 4 | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lung carcinoma cell type unspecified stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Renal cell carcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Thyroid cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0
Encephalitis (Nervous system disorders) | 0 | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 0 | 0
Ischaemic cerebral infarction (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1
Mental status changes (Psychiatric disorders) | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1
Renal colic (Renal and urinary disorders) | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Aortic stenosis (Vascular disorders) | 1 | 0 | 0
Capillary leak syndrome (Vascular disorders) | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0
Shock (Vascular disorders) | 1 | 0 | 0
Thrombophlebitis superficial (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Epoetin Alfa (80,000 Units) (N=75) | Epoetin Alfa (120,000 Units) (N=77) | Darbepoetin Alfa (500 Mcg) (N=75)
Anaemia (Blood and lymphatic system disorders) | 3 | 4 | 3
Neutropenia (Blood and lymphatic system disorders) | 12 | 17 | 14
Thrombocytopenia (Blood and lymphatic system disorders) | 7 | 8 | 7
Abdominal pain (Gastrointestinal disorders) | 7 | 5 | 5
Constipation (Gastrointestinal disorders) | 7 | 7 | 7
Diarrhoea (Gastrointestinal disorders) | 13 | 11 | 10
Nausea (Gastrointestinal disorders) | 11 | 12 | 9
Vomiting (Gastrointestinal disorders) | 7 | 9 | 8
Asthenia (General disorders) | 7 | 4 | 7
Fatigue (General disorders) | 15 | 15 | 16
Oedema peripheral (General disorders) | 8 | 6 | 6
Pain (General disorders) | 2 | 5 | 2
Pyrexia (General disorders) | 8 | 7 | 9
Sinusitis (Infections and infestations) | 0 | 4 | 4
Upper respiratory tract infection (Infections and infestations) | 0 | 5 | 1
Urinary tract infection (Infections and infestations) | 2 | 7 | 6
Weight decreased (Investigations) | 7 | 4 | 2
Anorexia (Metabolism and nutrition disorders) | 12 | 6 | 5
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 4
Dehydration (Metabolism and nutrition disorders) | 5 | 6 | 6
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 6 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 4 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 4 | 3
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 4 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 1 | 5
Dizziness (Nervous system disorders) | 7 | 5 | 6
Dysgeusia (Nervous system disorders) | 1 | 4 | 2
Headache (Nervous system disorders) | 4 | 4 | 4
Neuropathy (Nervous system disorders) | 3 | 7 | 4
Anxiety (Psychiatric disorders) | 3 | 5 | 2
Depression (Psychiatric disorders) | 3 | 3 | 4
Insomnia (Psychiatric disorders) | 3 | 7 | 7
Haematuria (Renal and urinary disorders) | 1 | 0 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 10
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 7 | 7
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 5 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 4 | 2
Rash (Skin and subcutaneous tissue disorders) | 4 | 4 | 7
Hypotension (Vascular disorders) | 2 | 6 | 4

LIMITATIONS AND CAVEATS:
Due to the significantly reduced power (stopped prematurely when 235 patients enrolled), all protocol-specified hypothesis tests were not performed. Instead, desriptive statistics were presented for each of the endpoints by treatment group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days